CLINICAL TRIAL: NCT01787500
Title: A Phase I Trial of Vemurafenib in Combination With Cetuximab and Irinotecan in Patients With BRAF V600 Mutant Advanced Solid Malignancies
Brief Title: Vemurafenib, Cetuximab, and Irinotecan Hydrochloride in Treating Patients With Solid Tumors That Are Metastatic or That Cannot Be Removed by Surgery
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0748; NCI-2013-00541 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2012-0748 (Other: M D Anderson Cancer Center); P30CA016672 (NIH); R01CA187238 (NIH)
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: BRAF NP_004324.2:p.V600X; KRAS wt Allele; Metastatic Malignant Solid Neoplasm; Stage IV Colorectal Cancer AJCC v7; Stage IVA Colorectal Cancer AJCC v7; Stage IVB Colorectal Cancer AJCC v7; Unresectable Solid Neoplasm
MeSH Terms: conditions — Noonan syndrome 3; Neoplasm Metastasis; Colorectal Neoplasms | interventions — Cetuximab; Irinotecan; Vemurafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (vemurafenib, cetuximab, irinotecan hydrochloride) (Experimental): Patients receive vemurafenib PO BID on days 1-14, cetuximab IV over 90 minutes, and irinotecan hydrochloride IV over 90 minutes on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Cetuximab; Drug: Irinotecan Hydrochloride; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Vemurafenib

INTERVENTIONS:
Biological: Cetuximab — Given IV
  Other Names: Cetuximab Biosimilar CMAB009; Chimeric Anti-EGFR Monoclonal Antibody; Chimeric MoAb C225; Chimeric Monoclonal Antibody C225; Erbitux; IMC-C225
Drug: Irinotecan Hydrochloride — Given IV
  Other Names: Campto; Camptosar; Camptothecin 11; Camptothecin-11; CPT 11; CPT-11; Irinomedac; U-101440E
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Vemurafenib — Given PO
  Other Names: BRAF (V600E) kinase inhibitor RO5185426; BRAF(V600E) Kinase Inhibitor RO5185426; PLX-4032; PLX4032; RG 7204; RG7204; RO 5185426; Zelboraf

SUMMARY:
This phase I trial studies the side effects and best dose of vemurafenib when given together with cetuximab and irinotecan hydrochloride in treating patients with solid tumors that have spread to other parts of the body or cannot be removed by surgery. Vemurafenib and irinotecan hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as cetuximab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving vemurafenib with cetuximab and irinotecan hydrochloride may be a better treatment for solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To define the maximum tolerated dose (MTD) of vemurafenib when used in combination with cetuximab and irinotecan (irinotecan hydrochloride).

II. To define the safety profile of this combination. III. To determine the antitumor activity of this combination specifically in patients with advanced solid malignancies with positive v-raf murine sarcoma viral oncogene homolog B (BRAF) (V600)/negative Kirsten rat sarcoma viral oncogene homolog (K-RAS) mutation. (Part II-expanded cohort) IV. To determine the antitumor activity of this combination in patients with metastatic colorectal cancer with positive BRAF (V600)/negative K-RAS mutation. (Part II-expanded cohort)

SECONDARY OBJECTIVES:

I. To evaluate clinical response signals of the combination. II. To assess the pharmacokinetic (PK) and pharmacodynamic (PD) profile of the combination.

OUTLINE: This is a dose-escalation study of vemurafenib.

Patients receive vemurafenib orally (PO) twice daily (BID) on days 1-14, cetuximab intravenously (IV) over 90 minutes, and irinotecan hydrochloride IV over 90 minutes on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed malignancy that is metastatic or unresectable
* Cancers with positive BRAF V600 mutation detected by a Clinical Laboratory Improvement Act (CLIA)-certified laboratory
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Life expectancy of greater than 3 months
* Patients must have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
* Patients must have a K-RAS wild-type (WT) tumor
* Absolute neutrophils count >= 1500/mcl (within 14 days)
* Platelets >= 100000/mcl (within 14 days)
* Hemoglobin (Hb) >= 9 mg/dl (within 14 days)
* Total bilirubin =< 1.5 mg/dl (within 14 days)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 5 x upper limit of normal if liver metastases present; otherwise, then =< 2.5 x upper limit (within 14 days)
* Estimated creatinine clearance by Cockcroft-Gault equation > 30 mL/min (within 14 days)
* Current treatment may cause harm to the developing human fetus; for this reason women of child-bearing age must have a negative pregnancy test at screening and both women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation, and for 6 months after last dose; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Signed informed consent approved by the Institutional Review Board prior to patient entry
* Expansion cohort: We propose a final expansion cohort for this study in a subset of interest utilizing the recommended dosing of combination; this cohort will include patients harboring characteristics that may predict response of combination or with clinical features that proved to derive most benefit of the study combination during preclinical studies; cancers with positive BRAF (V600) mutation detected by a CLIA-certified laboratory

Exclusion Criteria:

* Patient receiving any concurrent chemotherapy
* Concurrent severe and/or uncontrolled medical disease including, but not limited to, ongoing or active infection requiring intravenous antibiotics, bowel obstruction
* Symptomatic congestive heart failure (New York Heart Association [NYHA] class III or IV), or unstable angina pectoris
* Patients who have had a myocardial infarction, transient ischemic attack, unstable angina, or cardiovascular symptoms (CVS) within 6 months before treatment
* Presence of symptomatic pleural and/or pericardial effusion not appropriately treated
* Prolonged corrected QT (QTc) interval (>= 450 msec) as calculated by Bazett's formula, or patients with a history of congenital long QT syndrome or uncorrectable electrolyte abnormalities
* Medical and/or psychiatric problems of sufficient severity to limit full compliance with the study or expose patients to undue risk
* Known anaphylactic or severe hypersensitivity to the study drugs or their analogs
* Patient has failed to recover from any prior surgery within 4 weeks of study entry
* Patient is pregnant, lactating, or breastfeeding
* Patient has had any treatment specific for tumor control within 3 weeks of dosing with investigational drugs and cytotoxic agents, or within 2 weeks of cytotoxic agent given weekly, or within 6 weeks of nitrosoureas or mitomycin C, or within 5 half-lives of biological targeted agents with half-lives and pharmacodynamic effects lasting less than 5 days
* Patient is not able to swallow oral medication
* Patients receiving any medications or substances that are strong inhibitors or inducers of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) complex are ineligible
* Patients with known K-RAS mutant (codon 12 or 13) detected by a Food and Drug Administration (FDA)-approved test in a CLIA-certified laboratory
* Patients with BRAF WT cancers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2013-02-15 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of vemurafenib defined as the highest dose studied in which the incidence of dose limiting toxicity was less than 33% as graded by the National Cancer Institute Common Toxicity Criteria version 4.0 | Up to 4 weeks
  Descriptive statistics will be provided on the grade and type of toxicity by dose level.

CONTACTS AND LOCATIONS:
Overall Officials: David S Hong, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Hong DS, Morris VK, El Osta B, Sorokin AV, Janku F, Fu S, Overman MJ, Piha-Paul S, Subbiah V, Kee B, Tsimberidou AM, Fogelman D, Bellido J, Shureiqi I, Huang H, Atkins J, Tarcic G, Sommer N, Lanman R, Meric-Bernstam F, Kopetz S. Phase IB Study of Vemurafenib in Combination with Irinotecan and Cetuximab in Patients with Metastatic Colorectal Cancer with BRAFV600E Mutation. Cancer Discov. 2016 Dec;6(12):1352-1365. doi: 10.1158/2159-8290.CD-16-0050. Epub 2016 Oct 11. PMID 27729313
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org